CLINICAL TRIAL: NCT01450007
Title: Perineural Versus Systemic Dexamethasone as an Analgesic Adjunct to Ultrasound-Guided Ropivacaine Interscalene Blockade in Arthroscopic Rotator Cuff Repair
Brief Title: Ropivacaine Block Alone or With Perineural or Systemic Dexamethasone for Pain in Shoulder Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David Rosenfeld, Assistant Professor of Anesthesiology, College of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 11-001266
Record Dates: First submitted 2011-10-07; First posted 2011-10-10 (Estimated); Results first posted 2016-05-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-05

CONDITIONS: Shoulder Injury
Keywords: Pain blockade; Ropivacaine; Dexamethasone
MeSH Terms: conditions — Shoulder Injuries | interventions — Ropivacaine; Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dexamethasone block (Experimental): Blockade with 25 ml ropivacaine 0.5% mixed with 8 mg dexamethasone (0.8 ml), and 5 ml intravenous normal saline
  Interventions: Drug: Ropivacaine; Drug: Dexamethasone; Drug: Normal saline
- Dexamethasone IV (Active Comparator): Blockade with 25 ml ropivacaine 0.5% mixed with 0.8 ml normal saline, and intravenous 8 mg dexamethasone (0.8 ml dexamethasone, 4.2 ml saline) to total volume of 5 ml
  Interventions: Drug: Ropivacaine; Drug: Dexamethasone; Drug: Normal saline
- Placebo (Placebo Comparator): Blockade with 25 ml ropivacaine 0.5% mixed with 0.8 ml normal saline, and 5 ml intravenous normal saline
  Interventions: Drug: Ropivacaine; Drug: Normal saline

INTERVENTIONS:
Drug: Ropivacaine — 25 ml ropivacaine 0.5%
  Other Names: Naropin
Drug: Dexamethasone — 8 mg dexamethasone (perineural)
  Arms: Dexamethasone block
Drug: Dexamethasone — 8 mg dexamethasone (0.8 ml dexamethasone, 4.2 ml saline) to total volume of 5 ml (intravenous)
  Arms: Dexamethasone IV
Drug: Normal saline — 5 ml normal saline (intravenous)
  Arms: Dexamethasone block; Placebo
Drug: Normal saline — 0.8 ml normal saline (perineural)
  Arms: Dexamethasone IV; Placebo

SUMMARY:
Pre-operative perineural injection of dexamethasone mixed with local anesthetic in peripheral nerve blockade for orthopedic surgery has been shown to prolong the length of analgesia, improve visual analog pain scores, decrease post-operative opioid use, and decrease post-operative nausea. No study has been published to determine if this effect is a result of systemic absorption of dexamethasone or is a local effect of the drug on neuronal activity at the injection site. This study is a prospective, randomized, double-blind, controlled study to compare pain block with (1) ropivacaine and saline plus intravenous saline vs (2) ropivacaine and dexamethasone plus intravenous saline vs (3) ropivacaine and saline plus intravenous dexamethasone. Patients will be recruited sequentially and assigned to the three groups at random in equal ratios. The hypothesis is that dexamethasone injected perineurally in combination with ropivacaine for interscalene brachial plexus block will yield longer duration of sensory blockade as compared to ropivacaine alone without intravenous or perineural dexamethasone and as compared to ropivacaine and intravenous dexamethasone. This result will suggest that the effect of dexamethasone is a result of direct neuronal activity at the injection site versus systemic absorption.

ELIGIBILITY:
Inclusion criteria:

1. Patients undergoing elective shoulder surgery by one of two surgeons highly experienced in the procedure.
2. Patients are either: Opioid naïve; or Have not taken opiates for one month prior to surgery (tramadol is permissible).
3. Patients have an American Society of Anesthesiology physical status I-III.

Exclusion criteria:

1. Females who are pregnant.
2. Patients who are taking chronic daily opiates for one month prior to surgery except tramadol.
3. Diabetic patients.
4. Patients with creatinine above 1.1mg/dL for females and above 1.3mg/dL for males.
5. Patients with contralateral pneumothorax or diaphragmatic paralysis.
6. Patients with coagulopathy.
7. Patients with clinically significant previous nerve injury in surgical extremity.
8. Patients with an allergy to NSAIDs.
9. Patients who are refusing a block.
10. Patients with a contraindication to ropivacaine, dexamethasone, or interscalene block due to other medical condition such as severe chronic obstructive pulmonary disease (COPD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-05; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Rosenfeld, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rosenfeld DM, Ivancic MG, Hattrup SJ, Renfree KJ, Watkins AR, Hentz JG, Gorlin AW, Spiro JA, Trentman TL. Perineural versus intravenous dexamethasone as adjuncts to local anaesthetic brachial plexus block for shoulder surgery. Anaesthesia. 2016 Apr;71(4):380-8. doi: 10.1111/anae.13409. Epub 2016 Feb 22. PMID 26899862

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Mayo Clinic in Arizona from June 2012 to September 2014.
Pre-assignment Details: 238 patients were screened; of these 41 were excluded because they did not meet inclusion criteria, and 67 were excluded because they declined to be in the study.
Period: Overall Study
Arm/Group | Dexamethasone Block | Dexamethasone IV | Placebo
Started | 44 | 42 | 44
Completed | 42 | 37 | 41
Not Completed | 2 | 5 | 3
Not completed — Late exclusion before treatment | 2 | 3 | 2
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone Block | Dexamethasone IV | Placebo | Total
Number analyzed (Participants) | 42 | 37 | 41 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] — Baseline measures were provided for participants who completed the study.
  years | 67.5 (12.7) | 68.4 (7.7) | 62.7 (11.3) | 66.14 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 21 | 45
  Male | 29 | 26 | 20 | 75
Region of Enrollment [Number; unit: participants]
  United States | 42 | 37 | 41 | 120

OUTCOME MEASURES:

1. Primary Outcome: Duration of Sensory Blockade
Description: Duration from time of block until complete resolution of sensory blockade in the shoulder is recorded in minutes by patient report.
Time Frame: Within 48 hours
Population: Patients will be included in the primary analysis on the basis of intention to treat.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dexamethasone Block | Dexamethasone IV | Placebo
Number analyzed (Participants) | 42 | 37 | 41
hours | 16.9 (5.2) | 18.2 (6.4) | 13.8 (3.8)
Statistical Analysis 1: Comparison: Dexamethasone Block vs Dexamethasone IV; Test type: Superiority or Other; p = 0.001, ANOVA

2. Secondary Outcome: Post Operative Opioid Dose at 24 Hours
Time Frame: approximately 24 hours after surgery
Population: The number of participants analyzed is different from the number of participants in each arm who completed the trial because data were not available for 1 participant in the Dexamethasone IV group and 1 participant in the placebo group.
Measure: Mean (Standard Deviation); unit: mg morphine equivalents
Arm/Group | Dexamethasone Block | Dexamethasone IV | Placebo
Number analyzed (Participants) | 42 | 36 | 40
mg morphine equivalents | 12.2 (9.3) | 17.1 (15.9) | 24.1 (14.3)
Statistical Analysis 1: Comparison: Dexamethasone Block vs Dexamethasone IV vs Placebo; Test type: Superiority or Other; p = 0.001, ANOVA

3. Secondary Outcome: Time Until First Dose of Analgesic
Time Frame: Approximately 10 hours after surgery
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dexamethasone Block | Dexamethasone IV | Placebo
Number analyzed (Participants) | 42 | 36 | 40
hours | 8.4 (5.6) | 9.2 (5.6) | 8.4 (4.8)
Statistical Analysis 1: Comparison: Dexamethasone Block vs Dexamethasone IV vs Placebo; Test type: Superiority or Other; p = 0.76, ANOVA

4. Secondary Outcome: Patient Satisfaction With Pain Control
Description: Pain was rated on a visual analogue scale with 0 = no pain, 3=mild pain, 5=moderate pain, 7=moderate to severe pain, and 10=severe pain.
Time Frame: 24 hours, 48 hours, 1 week
Population: Patients analyzed for each category varied see explanations per row (time point): (n=dexamethasone block, dexamethasone IV, placebo).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexamethasone Block | Dexamethasone IV | Placebo
Number analyzed (Participants) | 42 | 37 | 41
units on a scale
  24 hours (n=34, 28, 37) | 7.8 (2.7) | 7.9 (2.6) | 7.3 (2.8)
  48 hours (n=42, 37, 41) | 8.4 (2.2) | 8.7 (2.0) | 7.6 (2.9)
  1 week (n=42, 36, 41) | 9.1 (1.2) | 8.8 (1.7) | 8.4 (2.4)
Statistical Analysis 1: Comparison: Dexamethasone Block vs Dexamethasone IV vs Placebo; Comparison between the 3 groups for pain scores at 24 hours; Test type: Superiority or Other; p = 0.61, Kruskal-Wallis
Statistical Analysis 2: Comparison: Dexamethasone Block vs Dexamethasone IV vs Placebo; Comparison between the 3 groups for pain scores at 48 hours; Test type: Superiority or Other; p = 0.13, Kruskal-Wallis
Statistical Analysis 3: Comparison: Dexamethasone Block vs Dexamethasone IV vs Placebo; Comparison between the 3 groups for pain scores at 1 week; Test type: Superiority or Other; p = 0.25, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: One week
Arm/Group | Dexamethasone Block | Dexamethasone IV | Placebo
Serious Adverse Events (participants affected / at risk) | 0/42 | 3/37 | 1/41
Other Adverse Events (participants affected / at risk) | 8/42 | 2/37 | 5/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone Block (N=42) | Dexamethasone IV (N=37) | Placebo (N=41)
Hospital admission for fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hospital admission for bowel infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Motor vehicle accident with fractured sternum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone Block (N=42) | Dexamethasone IV (N=37) | Placebo (N=41)
Skin rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
10 lb fluid weight within 24 hours (General disorders) | 1 (1) | 0 (0) | 0 (0) — Resolved without issue
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ER for nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fainting (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Frequent urination (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hoarse (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle soreness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Wrist, hand, and finger pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cranial nerve XII motor tongue (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Although it was designed to have 80% power at 120 patients, double this number would be required to detect very small differences (<10%) in the systemic and perineural groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes